CLINICAL TRIAL: NCT03436771
Title: Long-Term Follow-up Protocol for Subjects Treated With a CAR T-Cell Product on a Juno-Sponsored Clinical Trial
Brief Title: Long-term Follow-up Study for Patients Previously Treated With a Juno CAR T-Cell Product
Status: Terminated | Type: Observational
Why Stopped: Eligible subjects will be enrolled in Celgene's long-term follow-up protocol for subjects previously treated with a CAR T-cell product.
Sponsor: Juno Therapeutics, a Subsidiary of Celgene (Industry)
Responsible Party: Sponsor
Other Study IDs: LTFU001
Record Dates: First submitted 2018-02-12; First posted 2018-02-19 (Actual); Last update posted 2020-05-04 (Actual); Status verified 2020-04

CONDITIONS: Non Hodgkin Lymphoma; Multiple Myeloma; Chronic Lymphocytic Leukemia; Diffuse Large B Cell Lymphoma; Mantle Cell Lymphoma; Follicular Lymphoma
Keywords: long-term follow-up; chimeric antigen receptor (CAR) T cells; JCAR017; JCARH125
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Multiple Myeloma; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Mantle-Cell; Lymphoma, Follicular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Genomic DNA prepared from peripheral blood mononuclear cells
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- JCAR017-treated: Patients who received previous treatment with JCAR017
  Interventions: Genetic: JCAR017
- JCARH125-treated: Patients who received previous treatment with JCARH125
  Interventions: Genetic: JCARH125

INTERVENTIONS:
Genetic: JCAR017 — No drug is administered in this study. Patients who received JCAR017 in a previous trial will be evaluated in this trial for long-term safety and survival.
  Groups: JCAR017-treated
Genetic: JCARH125 — No drug is administered in this study. Patients who received JCARH125 in a previous trial will be evaluated in this trial for long-term safety and survival.
  Groups: JCARH125-treated

SUMMARY:
This study will provide long-term follow-up for patients who have received treatment with a Juno CAR T-cell product in a Juno-sponsored clinical trial. In this study, patients will be followed for up to 15 years after their last dose of Juno CAR T cells for evaluation of delayed adverse events, presence of persisting CAR T-cell vector sequences, presence of replication-competent retrovirus (RCR) or lentivirus (RCL), and survival.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have received at least one dose of a Juno CAR T-cell product (listed above) in a Juno-sponsored clinical trial
* Patients who have provided informed consent for the long-term follow-up study

Exclusion Criteria:

* None. All patients who have previously received treatment with a Juno CAR T-cell product are eligible for this long-term follow-up study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients previously treated with a Juno CAR T-cell product on a Juno-sponsored clinical trial
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2018-02-19 (Actual); Primary Completion 2018-07-20 (Actual); Study Completion 2018-07-20 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with adverse events | 15 years from last treatment
Proportion of patients with detectable viral vector sequences | 15 years from last treatment
Proportion of patients with detectable RCR or RCL | 15 years from last treatment

SECONDARY OUTCOMES:
Overall survival | 15 years from last treatment
Progression-free survival | 15 years from last treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Garcia, MD, Study Director — Sponsor GmbH
Locations (2):
- United States (2):
  - City of Hope, Duarte, California
  - Massachusetts General Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No